CLINICAL TRIAL: NCT04931381
Title: A Prospective, Randomized, Controlled Trial of Chemotherapy for Advanced Pancreatic Cancer Based on Organoid Drug Sensitivity Test
Brief Title: Organoid-Guided Chemotherapy for Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Associated Professor at the Institute of Pancreatic Surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP09
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Organoid; Drug Sensitivity Test; Chemotherapy; Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid-Guided Chemotherapy (Experimental): The pancreatic cancer specimens are obtained from biopsy to be cultured for organoids. Then drug sensitivity is tested using organoid to obtain the sensitivity to the first-line drugs for pancreatic cancer (Gemcitabine, 5-fluorouracil, Paclitaxel, Oxaliplatin, Irinotecan). Patients will receive relatively sensitive chemotherapy regimen based on the test results. Chemotherapy should start within 1 months after biopsy, and be given at least 1 cycle.
  Interventions: Other: Chemotherapy guided by organoid drug sensitivity test
- Physician-decided Chemotherapy (No Intervention): The pancreatic cancer specimens are obtained from biopsy to be cultured for organoids. Then drug sensitivity is tested using organoid to obtain the sensitivity to the first-line drugs for pancreatic cancer (Gemcitabine, 5-fluorouracil, Paclitaxel, Oxaliplatin, Irinotecan). Physician will decide the the adjuvant chemotherapy regimen, according to National Comprehensive Cancer Network (NCCN) guideline for pancreatic ductal adenocarcinoma. And they don't know the drug sensitivity test results. Chemotherapy should start within 1 months after biopsy, and be given at least 1 cycle.

INTERVENTIONS:
Other: Chemotherapy guided by organoid drug sensitivity test — Chemotherapy guided by organoid will be given to advanced pancreatic cancer patients.
  Arms: Organoid-Guided Chemotherapy

SUMMARY:
The purpose of this study is to explore whether chemotherapy regimens guided by organoid drug sensitivity test can improve the outcomes of advanced pancreatic cancer. At the same time, this study will evaluate the successful stablishment rate of organoid from biopsy tissue , and explore the concordance between drug sensitivity test results and patients' treatment response.

DETAILED DESCRIPTION:
The poor prognosis of pancreatic cancer is not just because of the high malignancy of the tumor itself, but also its poor response to chemotherapy. At present, patient's drug-sensitivity is assessed by progression time after treatment. Therefore, it is difficult to judge a patient's sensitivity to a drug before chemotherapy. Organoid is a new tumor model, which has the potential to test the drug sensitivity before chemotherapy.

Our center's previous experience has shown that the success rate of pancreatic cancer organoid culture is 77.6%. The previous research has confirmed that pancreatic cancer organoid was highly consistent with the original tissue in terms of genomics and histomorphology. More importantly, the investigators have tested the five first-line drug-sensitivity in 39 pancreatic cancer organoids, and compared the test results with the clinical treatment response of these patients, confirming that organoid can accurately evaluate the chemotherapy drug-sensitivity.

This is a single-center, prospective, open-label, randomized, controlled clinical trial, designed to explore whether chemotherapy regimens guided by organoid drug sensitivity test can improve outcomes in advanced pancreatic cancer patients. At the same time, the consistency between the drug sensitivity test results and the treatment response of patients will be analyzed. Also, the radiosensitivity of organoids will be tested, and be compared with the patients' response to radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old and ≤80 years old.
* Histologically or cytologically confirmed local advanced/metastatic pancreas adenocarcinoma.
* Eligible histologic variants include adenocarcinoma or variants to include mucinous adenocarcinoma or adenosquamous carcinoma.
* Patient must have a tumor lesion that is amenable to a core needle biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of greater than 90 days, as judged by the investigator.
* Routine blood test: absolute neutrophil count>1500/mm3, platelet>100000/mm3.
* Normal liver function: serum total bilirubin≤2.0mg/dl, alanine aminotransferase (ALT) and aspertate aminotransferase (AST) <2.5 times of the upper limit of normal value.
* Normal kidney function: serum creatinine<1.5 times of the upper limit of normal value or creatinine clearance rate>45ml/min.
* The pancreatic cancer organoid were cultured successfully.
* No severe comorbidities.

Exclusion Criteria:

* Patients with poor condition can not tolerate chemotherapy and targeted therapy.
* Impaired organ functions: heart failure (New York Heart Association III-IV), coronary heart disease, myocardial infarction within 6 months, severe cardiac arrhythmia and respiratory failure.
* Patients diagnosed with other cancer within 5 years.
* Patients who are pregnant or breastfeeding.
* Patients enrolled in other clinical trials or incompliant of regular follow up.
* Patients who did not provide an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
6-month disease control rate | 6 months
  Percentage of patient's measurable disease who have achieved either complete response (CR) , partial response (PR) or stable disease (SD) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression free time | 1-2 years
  Time from the date of randomization to progression based on the radiology assessment of response using RECIST v1.1, or death, whichever is earlier.
Overall survival time | 1-2 years
  The time from the date of randomization to the date of death for any cause. Patients will be followed until their date of death or until final database closure. Patients who are lost-to-follow-up or are alive at the time of analysis will be censored at the time they were last known to be alive or at the date of event cut-off for Overall survival (OS) analysis.
The successful establishment rate of organoids | 1-2 years
  The rate of organoid successfully cultured in all the samples collected.
Concordance between drug sensitivity test results and patients' treatment response (descriptive statistics). | 1-2 years
  To assess the accuracy of drug sensitivity test in both group. The number of patients with correct prediction of treatment response by organoid drug-sensitivity test divided by the number of patients underwent chemotherapy
Concordance between radiosensitivity test results and patients' treatment response (descriptive statistics). | 1-2 years
  To assess the accuracy of radiosensitivity test in both group. The number of patients with correct prediction of treatment response by organoid radiosensitivity test divided by the number of patients underwent radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, M.D., Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No